CLINICAL TRIAL: NCT05821621
Title: Efficacy and Safety of Cashew Nut Oral Immunotherapy in Children
Acronym: CAJESITO2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Amandine DIVARET-CHAUVEAU, PhD, Central Hospital, Nancy, France
Other Study IDs: 2022PI216
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Food Allergy in Children
Keywords: Cashew nut allergy; Food allergen immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cashew nut allergy: Inclusion criteria:
  * Patients under 18 years of age with a proven allergy to cashew nut and followed in the pediatric allergology unit of Nancy University Hospital.
  * Patients having received oral cashew immunotherapy for at least 18 months at 28/02/2023
  Non-inclusion criteria:
  * Patients who have received oral cashew immunotherapy for less than 18 months.
  * Patients lost to follow-up for more than 3 years (last consultation in 2020 or earlier)
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — observational study : there is no intervention

SUMMARY:
Allergy to nuts (cashew, pistachio, walnut, exotic nuts) is a frequent allergy in children, with a prevalence of up to 4.9% of the population and a low resolution rate (9%). Among the nut allergies, cashew nut allergy is one of the most frequent in Northern Europe: in France 41% of children allergic to nuts are sensitized to cashew nuts. Moreover, cashew nut allergy is associated with severe reactions that can be lethal in both adults and children. These reactions may even be more severe than those observed with peanuts, with more frequent respiratory and cardiovascular impairment. We note reactions for even limited contacts (cutaneous or mucous) and low reactogenic thresholds. However, the only recommendation for management at present is avoidance. The stakes of oral immunotherapy protocols cashew would be similar to those for peanut immunotherapy: to limit reactions in case of accidental intake, increase the reactogenic threshold and thus improve the quality of life of allergic patients.

To date, only one study has focused on the efficacy and tolerance of cashew immunotherapy : the prospective NUT CRACKER study conducted on 50 children aged 4 years or older with cashew nut allergy between 2016 and 2019, reports a good efficacy of immunotherapy on increasing threshold for cashew nut but also for pistachio and walnut, when there was a cross-over allergy. While the tolerance was similar to other immunotherapy protocols for the other foods.

The objectives of part 2 of the CAJESITO study are (i) to evaluate the tolerance of oral cashew nut immunotherapy, by describing the frequency and severity of allergic reactions during oral cashew immunotherapy and (ii) to identify risk factors for severe risk factors for severe allergic reactions during oral cashew immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 18 years of age with a known allergy to cashew nuts cashew nut allergy and followed in the pediatric allergology unit of Nancy University Hospital.
* Patients who have received oral cashew immunotherapy for at least 18 months at 28/02/2023

Exclusion Criteria:

* Patients who have received oral cashew immunotherapy for less than for less than 18 months.
* Patients lost to follow-up for more than 3 years (last visit in 2020 or earlier)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Observational, longitudinal and monocentric epidemiological study carried out in the pediatric allergology department of the Nancy University Hospital.
  Data collection will be carried out retrospectively. The study does not foresee any new collection of health data. No follow-up will be necessary for the patients of the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-04-17 (Estimated); Primary Completion 2023-04-17 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Safety | during the dose escalation phase and during 6 months of maintenance
  To evaluate the safety of oral cashew immunotherapy during the dose escalation phase and during the maintenance phase : Frequency of occurrence of at least one allergic reaction during the dose escalation phase and during the first 6 months of maintenance

SECONDARY OUTCOMES:
Frequency of allergic reaction | during the dose escalation and maintenance phases : first 6 months, 1st year, 2nd year, 3rd year
  To assess the frequency of allergic reactions reactions during the dose escalation and maintenance phases : Frequency of allergic reactions during the dose-escalation and maintenance phases (first 6 months, 1st year, 2nd year, 3rd year)
Describe the severity of allergic reactions | during the dose escalation and maintenance phases (first 6 months, 1st year, 2nd year, 3rd year)
  Describe the severity of allergic reactions during the dose escalation and maintenance phases : Severity of allergic reactions during the dose escalation and during the maintenance phase (first 6 months, 1st year, 2nd year, 3rd year)
Predictive factors of severe allergic reactions | during cashew nut immunotherapy
  To identify predictive factors of severe allergic reactions during cashew nut immunotherapy : Predictive factors for the occurrence of severe allergic reactions (age at initiation, atcd of severe allergic reaction, initial threshold, asthma, other food allergy, atopic dermatitis, allergic rhinitis, initial specific IgE levels, ratio IgE rAna o3/cashew ratio)
Factors associated with severe allergic reactions | during cashew nut immunotherapy
  identify the factors (during the protocol) associated with severe allergic reactions (cofactor, poor compliance...) : Factors associated with the occurrence of severe allergic reactions (bad compliance, fasting, pollen peak, infection, asthma imbalance, effort, excitement, medication...)
Immunotherapy discontinuation | during cashew nut immunotherapy
  Evaluate the frequency of immunotherapy discontinuation and describe its causes

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalo-Universitaire de Nancy, Vandœuvre-lès-Nancy, France